CLINICAL TRIAL: NCT04768829
Title: Antifungal Potential of Moringa Olifera-loaded Nanoparticles Against Otomycosis; Preparation, Characterization, and Clinical Evaluation
Brief Title: Antifungal Potential of Moringa Olifera Against Otomycosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Deraya University (Other)
Collaborators: Minia University (Other)
Responsible Party: Principal Investigator, Soad Ali, principle investigator, Deraya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S85Motic
Record Dates: First submitted 2021-02-18; First posted 2021-02-24 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis | interventions — Urea

STUDY DESIGN:
Intervention Model Description: moringa extract ear drops
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Active Comparator): Nystatin ear drops formulations prepared as intervention except for the addition of Moringa prepared using biodegradable polymers in aseptic condition and tested for sensitivity
  Interventions: Drug: Ear Drop
- Moringa group (Experimental): Moringa ear drops prepared using biodegradable polymers in aseptic condition and tested for sensitivity
  Interventions: Drug: Moringa oleifera leaf 10mg/100ml

INTERVENTIONS:
Drug: Moringa oleifera leaf 10mg/100ml — ear drops
  Other Names: ear drops
  Arms: Moringa group
Drug: Ear Drop — plain ear drop formulation without moringa
  Arms: Placebo group

SUMMARY:
patients with Otomycosis were recognized by an ENT specialist. 20 patients were distributed randomly into two groups. The first group will be treated with Nystatin ear drops twice daily. The second group will be treated with Moringa ear drops. patients will be examined endoscopically by the ENT specialist. patient's swabs will be isolated and analyzed by ELISA.

DETAILED DESCRIPTION:
Inclusion criteria:

(1) Otomycosis .

Exclusion criteria:

1. tympanic membrane perforation;
2. concurrent immune suppression,
3. and concurrent bacterial infection.

ELIGIBILITY:
Inclusion Criteria:

1. Otomycosis
2. ear inflammation

Exclusion Criteria:

1. tympanic membrane perforation
2. concurrent immune suppression,
3. concurrent bacterial infection.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Number of participants recovered with clear endoscopic examination | one week
  Number of participants recovered with clear endoscopic examination
Identification of different microorganisms infected ear | up to 1 month
  Patients swabs (microorganisms concentration)

CONTACTS AND LOCATIONS:
Overall Officials: Soad A Mohamad, Principal Investigator — Deraya University
Locations (1):
- Soad A. Mohamad, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publication in peer-reviewed journals
Supporting Information: Study Protocol, SAP
Time Frame: year